CLINICAL TRIAL: NCT03239366
Title: A Double-blind, Randomized Placebo Controlled Study to Evaluate the Effect of BioK+ 50B® on Glycemic Control in a Type 2 Diabetes Population
Brief Title: A Study to Evaluate the Effect of BioK+ 50B® on Glycemic Control in a Type 2 Diabetes Population
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: Montreal Heart Institute (Other); The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ProbioHeart 2017.18
Record Dates: First submitted 2017-07-27; First posted 2017-08-04 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Type2 Diabetes
Keywords: T2D
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This study will evaluate the effects of Bio-K+50B® at a dosage of 100 billion (B) colony forming units (CFU) daily for 12 weeks in improving glycemic control in patients with Type 2 diabetes (T2D) population when compared to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double blind, randomized and placebo controlled. The clinical and operational teams from both MHI and BioK+ are blinded. Treatment codes will be available at the research pharmacy from the MHI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Active product 'BioK+ 100% probiotic: Bio-K+50B® probiotic will be administered orally for a period of 12 weeks. Dose: two (2) capsules of 50 billion (B) colony forming units (CFU) providing a dosage of 100 billion CFU per day
  Interventions: Other: BioK+ 100% probiotic
- Placebo arm (Placebo Comparator): Placebo product (without the 3 strains of bacterias) will be administered orally for a period of 12 weeks. Dose: Two (2) capsules of Placebo per day
  Interventions: Other: Placebo

INTERVENTIONS:
Other: BioK+ 100% probiotic — The active BioK+ product will include the 3 strains of Lactobacillus: L. acidophilus CL1285®, L. casei LBC80R® and L. rhamnosus CLR2®, representing the bacteria found in Bio-K+ probiotic capsules 50B®;
  Arms: Active arm
Other: Placebo — The placebo product will NOT include the 3 strains of Lactobacillus: L. acidophilus CL1285®, L. casei LBC80R® and L. rhamnosus CLR2®, representing the bacteria found in Bio-K+ probiotic capsules 50B®;
  Arms: Placebo arm

SUMMARY:
This study will be conducted at the Montreal Heart Institute and should involve 130 Type 2 diabetes subjects. Subjects will be randomized in a 1:1 ratio to receive either Bio-K+50B® probiotic capsules or a matching placebo.

DETAILED DESCRIPTION:
This is a phase 2 double-blind, randomized, single-center, placebo-controlled, parallel-group 12-week study of Bio-K+ probiotic 50B® in subjects diagnosed with Type 2 diabetes (T2D) and suboptimal glycemic control.

After providing informed consent and completion of screening baseline assessments, approximately 130 subjects will be randomized in a 1:1 ratio to receive either Bio-K+50B® probiotic or matching placebo. Subjects will take investigational product or placebo once daily orally for 12 weeks.

During the double-blind treatment period, subjects will complete a daily diary and will be contacted via telephone (at Week 4 and Week 8) for an assessment of adverse events, concomitant medications, diabetes management habits, collection of stool sample at home, diary revision and study product compliance. At visit 3 (Week 12; end of study visit) subjects will return to the study site for laboratory tests and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet ALL of the following inclusion criteria in order to be eligible for this study:

  1. Aged 18 years and older on the day of consent;
  2. T2D diagnosis according to Canadian diabetes guidelines[24] and treated with medication for this diagnosis;
  3. Suboptimal glycemic control, as evidenced by HbA1c >7%;
  4. Body Mass Index (BMI); greater than or equal to 25 and less than 40 kg/m2
  5. Subjects willing to maintain a stable diet and physical activity level throughout the study;
  6. Ability and willingness to give written informed consent and to comply with the requirements of the study.
  7. The subject is able to read and write English or French.

Exclusion Criteria:

* A patient who meets any of the following criteria will NOT be eligible to the study:

  1. Subjects unlikely to cooperate in the study;
  2. Legal incapacity or limited legal capacity;
  3. Women who are pregnant, planning to become pregnant during the study or breast-feeding. Women of childbearing potential must have a negative urine pregnancy test at screening. Women are considered not of childbearing potential if they:

     1. Have had a hysterectomy or tubal ligation prior to Visit 1.
     2. Are postmenopausal defined as no menses for 12 months or a Follicle-stimulating Hormone (FSH) level in the menopausal range.

     Women of childbearing potential must agree to use an effective method of birth control throughout the study. Acceptable means of birth control include: implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, diaphragm with spermicide, male or female condoms with spermicide or cervical cap, abstinence, or a sterile sexual partner.
  4. Participation in a drug or device trial within the previous 30 days (or within 5 half-lives of the investigational drug, or within the time legally required by local regulatory authorities, whichever is the longest) or participation in such trial considered, or patient already enrolled in the study. Participation to observation registries is allowed;
  5. Type 1 diabetes;
  6. Gestational diabetes;
  7. Diabetes secondary to:

     * Genetic defects of beta (β) cell function (Maturity-Onset Diabetes of the Young) or insulin action;
     * Diseases of the exocrine pancreas (pancreatitis, neoplasia, cystic fibrosis, hemochromatosis);
     * Endocrinopathies (Acromegaly, Cushing's syndrome, glucagonoma, pheochromocytome, hyperthyroidism);
     * Drugs (glucocorticoids, clozapine),
     * Infections (Congenital rubella, Cytomegalovirus, coxsackie);
     * Genetic syndromes associated with diabetes (Down's syndrome, Klinefleter's syndrome, Turner's syndrome);
  8. Subjects whose medication for glycemic control has been changed in the past 3 months or whose medication is likely to be changed during the conduct of the study;
  9. Chronic gastro-intestinal illness (e.g. Crohn's disease, ulcerative colitis, colon cancer);
  10. Prior abdominal surgery that, in the investigator's opinion, may confound study outcomes;
  11. Current treatment with nasogastric tube, ostomy, or parenteral nutrition;
  12. Immunodeficiency;
  13. Morbid obesity, as evidenced by Body Mass Index (BMI) ≥ 40;
  14. Eating disorder;
  15. Uncontrolled mental illness that could interfere with the conduct of the study;
  16. Known pancreatic disease, other than diabetes mellitus;
  17. Known severe renal disease (creatinine ≥200 micromoles per liter);
  18. Known moderate or severe liver disease (enzymes alanine transaminase (ALT) or aspartate transaminase (AST) > 3 times upper normal limit);
  19. Significant anemia defined as blood hemoglobin lower than 110 grams per liter (in males) or lower than 100 grams per liter (in females);
  20. History of alcohol, medication or drug abuse;
  21. History of smoking in the past 12 months;
  22. Daily consumption of prebiotics and/or probiotics;
  23. Daily consumption of fermented milk (more than 1 litre a day);
  24. Known allergies to any substance in the study product or placebo;
  25. Any serious disease likely to interfere with the conduct of the study or compromise subject safety;
  26. Life expectancy shorter than 6 months;
  27. Subjects requiring treatments which will not be tolerated in this study (refer to Appendix 2);
  28. Lactose intolerance or allergy to cow's milk protein;
  29. Any condition or therapy that the investigator believes might pose a risk to the patient or make participation in the study not in the patient's best interest; Chronic and regular usage of anti-inflammatory drugs and recent use (in the last three months) of oral antibiotics will not be tolerated in the context of this study because of their well-recognized modifying effect of the intestinal flora;
  30. Known heart failure and/or left ventricular ejection fraction less than 30%;
  31. Insulin therapy;
  32. Taking a natural health product that may affect blood glucose levels such as chromium, cinnamon bark, or bitter melon product.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c levels from baseline | 12 weeks
  The primary objective is to evaluate the effect of Bio-K+50B® on HbA1c level compared with placebo after 12 weeks of treatment in subjects with T2D and suboptimal glycemic control (HbA1c >7% at baseline).

SECONDARY OUTCOMES:
Evaluation of the effects of Bio-K+50B® as compared with placebo after 12 weeks of treatment on different biochemical markers: | 12 weeks
  The following biochemical markers will be measured:
  • Fasting blood glucose, lipid profile, high-sensitivity C-Reactive Protein (hs-CRP), creatinine, homeostatic model assessment insulin resistance (HOMA-IR) and fasting insulin.
Evaluation of the intestinal colonisation effects with the 2 capsules of Bio-K+50B® (dosage of 100 billions bacterias) as compared with placebo | 12 weeks
  Measurement of fecal concentrations of bacteria found in Bio-K+50B®: L. acidophilus CL 1285® + L. casei LBC80R® and L. rhamnosus CLR2®;
Evaluation of the safety profile of 2 capsules of Bio-K+50B® (dosage of 100 billions bacterias) | 12 weeks
  During the full course of the study, the investigator is responsible for the detection and documentation of events meeting the criteria and definition of an AE or a SAE.
  Abnormal laboratory findings (e.g. clinical chemistry, hematology, urinalysis) or other abnormal assessments (e.g. vital signs) that are judged by the investigator as clinically significant will be recorded as AEs or SAEs.
  A daily diary will be completed by the subject in order to assess overall diabetes management. The diary includes collection of information on symptoms of hypoglycaemia. In addition, information will be collected on gastrointestinal symptoms and any other new symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude Tardif, MD, Principal Investigator — Cardiologist at the MHI
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tonucci LB, Olbrich Dos Santos KM, Licursi de Oliveira L, Rocha Ribeiro SM, Duarte Martino HS. Clinical application of probiotics in type 2 diabetes mellitus: A randomized, double-blind, placebo-controlled study. Clin Nutr. 2017 Feb;36(1):85-92. doi: 10.1016/j.clnu.2015.11.011. Epub 2015 Dec 7. PMID 26732026
- [Result] Ferguson JF, Allayee H, Gerszten RE, Ideraabdullah F, Kris-Etherton PM, Ordovas JM, Rimm EB, Wang TJ, Bennett BJ; American Heart Association Council on Functional Genomics and Translational Biology, Council on Epidemiology and Prevention, and Stroke Council. Nutrigenomics, the Microbiome, and Gene-Environment Interactions: New Directions in Cardiovascular Disease Research, Prevention, and Treatment: A Scientific Statement From the American Heart Association. Circ Cardiovasc Genet. 2016 Jun;9(3):291-313. doi: 10.1161/HCG.0000000000000030. Epub 2016 Apr 19. PMID 27095829
- [Derived] Cuthill S, Muroke V, Dubois A, Dube MP, Guertin MC, Millette M, Tardif JC. Effect of probiotic supplementation on glycemic control in patients with type 2 diabetes: A randomized controlled trial. Clin Nutr ESPEN. 2025 Aug;68:148-152. doi: 10.1016/j.clnesp.2025.05.013. Epub 2025 May 7. PMID 40345656